CLINICAL TRIAL: NCT06124560
Title: An Oral Single-dose, Randomized, Balanced, Open-label, Two-sequence, Two-treatment, Two-period, Crossover Bioequivalence Study of Sitagliptin Hydrochloride / Metformin Hydrochloride Extended-release Film Coated Tablets 100 mg /1000 mg (FDC) of Galenicum Health S.L.U., Spain With That of JANUMET® XR (Sitagliptin Phosphate / Metformin Hydrochloride) Extended-release Coated Tablets 100 mg / 1000 mg (FDC) of Merck Sharp & Dohme Pharmaceuticals Ltd., Brazil in Healthy Adult Male and Female Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Sitagliptin Hydrochloride / Metformin Hydrochloride Extended-release Film Coated Tablets 100 mg /1000 mg (FDC) in Healthy Adult Male and Female Subjects Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galenicum Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AS/CJ/ENE-22/0005
Record Dates: First submitted 2023-07-25; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Bioequivalence; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (Experimental): After an overnight fasting of at least 10.00 hours prior to dosing, subjects were administered a single-dose of the reference product along with 250 mL of 20% glucose in water solution at room temperature.
  Interventions: Drug: Sitagliptin/Metformin HCl 100/1000 mg extended release film-coated tablet
- Test group (Experimental): After an overnight fasting of at least 10.00 hours prior to dosing, subjects were administered a single-dose of the test product along with 250 mL of 20% glucose in water solution at room temperature.
  Interventions: Drug: Sitagliptin/Metformin HCl 100/1000 mg extended release film-coated tablet

INTERVENTIONS:
Drug: Sitagliptin/Metformin HCl 100/1000 mg extended release film-coated tablet — The subjects randomly received single oral dose of Sitagliptin/Metformin HCl 100/1000 mg extended release film-coated tablet

SUMMARY:
The objective of this study was to evaluate and compare the bioavailability and therefore to assess the bioequivalence of two different formulations of sitagliptin/metformin extended release tablets after a single oral dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female subjects aged ≥ 18 and ≤ 55 years.
2. Subjects is a non-or ex-smoker.
3. With a weight ≥ 50.00 kg.
4. With a body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 27.0 kg/m2.
5. Found healthy according to the clinical laboratory results and physical examination
6. Have a normal 12-lead ECG and vital signs.
7. Have laboratory test results within the laboratory's stated normal range; if not within this range, they must lack of clinical significance as judged by the PI or responsible physician.
8. If the subject of the study is female and childbearing potential / fertile (a woman is considered fertile from first menstruation and until she becomes postmenopausal, or permanently sterile), and agrees to use ANY ONE of the following forms of effective contraception / birth control (but not limited to) from the time of enrollment into the study and until at least 7 days after the last study drug administration, as judged by the PI considering the pharmacology of IP(s):

   1. Established use of oral, transdermal, injected or subdermal implanted hormonal methods.
   2. Intrauterine device (IUD or intrauterine system (IUS).
   3. Barrier methods: e.g., diaphragm, cervical cap or condom (male or female condom).
   4. Spermicidal: e.g., spermicidal foam, sponges or film.
   5. Undergone bilateral tubectomy.
   6. Accept to remain abstinent: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception]

   Women who are postmenopausal (defined as female with no menses at least for the last 12 months without any medical cause) or permanently sterilized (e.g., undergone hysterectomy, bilateral salpingectomy or oophorectomy at least for the last 3 months).
9. If the subject of the study is male, he must be willing to use ANY ONE of the following forms of effective contraception / birth control (but not limited to) and willing not to donate sperm; from the time of enrollment into the study and until at least 7 days after the last study drug administration, as judged by the PI;

   1. Willing to remain abstinent: When this is in line with the preferred and usual lifestyle of the subject.
   2. Willing to use a male condom.
   3. Male sterilization (men who have had vasectomy, at least 3 months previous to drug administration).
10. Subject able to communicate effectively and voluntarily agreed to participate in this study by signing written informed consent after being informed sufficiently about study aspects like objectives, study procedures, characteristics of the investigational drug, expected adverse events.
11. Subject willing to adhere to protocol requirements as evidenced by signing the informed consent form approved by the REC & RC.

Exclusion Criteria:

1. Have any history of allergy or hypersensitivity to sitagliptin and metformin or to any of its metabolites/derivatives or related drugs or excipients.
2. Have a positive test result for HBs Ag or HCV Ab or HIV antibodies (types 1 and 2) or VDRL.
3. The study drug is contraindicated for medical reasons for the subject as per protocol section 3.7.
4. Have any history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, neurological or psychiatric disease or disorder (e.g., subjects with uncontrolled hypertension, phaeochromocytoma, carcinoid, thyrotoxicosis, bipolar depression, schizoaffective disorder and acute confusional states) as judged by the PI considering the pharmacology of IP(s).
5. Presence of gastrointestinal, hepatic or kidney disease, or surgery or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.

   Or Subjects with a history of gastrointestinal disorder or surgery which may affect the absorption of investigational drug.
6. Have history or presence of Corona Virus Disease (COVID-19) during the last 30 days prior to dosing of period 1.

   Or Have history of vaccination (any dose) for COVID-19 during the last 14 days prior to dosing of period 1.

   Or Any planned vaccination for COVID-19 during the study period.
7. Have history or presence of cancer.
8. Have a history or evidence of drug abuse or alcohol abuse.
9. Have a history of smoking cigarettes during the last 6 months prior to screening.
10. Have any history of gastrointestinal ulcers / bleeding.
11. Have difficulty in swallowing solid medications such as tablet.
12. Have a history or evidence of difficulty with donating blood.
13. Have clinically significant abnormal laboratory tests results.
14. Have a systolic blood pressure < 90 or > 140 mmHg or diastolic blood pressure is < 60 or > 90 mmHg
15. Have a pulse rate less than 60 bpm or greater than 100 bpm (lower range will be accepted up to 45 bpm in case of athlete).
16. Have used any prescribed medication during the last 14 days preceding the first dosing, or use OTC, herbal products during the last 7 days or use medicinal enzyme inhibitors / inducers during 30 days preceding the first dosing.
17. Have participated in a drug research study the last 3 months or donated blood within the last 3 months.
18. Have a positive result for the alcohol test (breath / saliva) or drugs of abuse test [Cannabinoids (Marijuana/Tetrahydrocannabinol-THC), Cocaine, Opiates/Morphine, Amphetamine, Methamphetamine and Benzodiazepines] performed during screening.
19. Female subject, who is currently breast feeding or a who is pregnant or who is likely to become pregnant during the study.
20. Female subject has a positive pregnancy test result.
21. Unwillingness or inability to comply with the instructions on the restrictions and/or study procedures described in the Protocol.
22. If the PI considers, for any reason, that the volunteer is not a suitable candidate to receive the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 48 hours
  Evaluation of Area Under Plasma Concentration-Time Curve from Time Zero to the Last Measurable Concentration
Area under the plasma concentration versus time curve (AUC) 0-inf (Metformin only) | 48 hours
  Area Under Plasma Concentration-Time Curve from Time 0 to Infinite

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | 1 week
  To evaluate the safety and tolerability of a single oral dose of Sitagliptin /Metformin extended-release film coated tablets 100 mg /1000 mg (FDC) under fasting conditions

CONTACTS AND LOCATIONS:
Overall Officials: María Elena Cedano Limón, Principal Investigator — Avant Santé Research Center S.A. de C.V.
Locations (1):
- Avant Santé Research Center S.A. de C.V., San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No